CLINICAL TRIAL: NCT07110766
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase Ib Clinical Study to Evaluate the Efficacy and Safety of Small Molecule MDR-001 Tablets Administered Orally for 12 Weeks Treatment in Overweight or Obesity Participants
Brief Title: Phase Ib Clinical Study on the Efficacy and Safety of MDR-001 in Patients Who Are Obesity or Overweight
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MindRank AI Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDR-001-CN-04
Record Dates: First submitted 2025-07-23; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDR-001 (Experimental): MDR-001 Administered orally
  Interventions: Drug: MDR-001
- Placebo (Experimental): Administered orally placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDR-001 — Oral administration of small molecule MDR-001 tablets
  Arms: MDR-001
Drug: Placebo — Administered orally placebo
  Arms: Placebo

SUMMARY:
This is a 12 weeks, multicenter, randomized, double-blind, placebo, parallel-controlled Phase Ib trail comparing the efficacy and safety of MDR-001 tablet versus placebo as an adjunct to a reduced calorie diet and increased physical activity in subjects with overweight or obesity, and to explore the optimal dose selection to support the subsequent Pivotal trial.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate in this study.
* Chinese male or female participants who are aged 18-65 (inclusive) years at the time of signing the ICF.
* Participants who are obesity (BMI ≥ 28.0 kg/m2), or overweight (24.0 kg/m2 ≤ BMI < 28.0 kg/m2) with at least one of the following weight-related comorbidities at screening:

  1. Pre-diabetes: 6.1 mmol/L (110 mg/dL) ≤ FPG < 7.0 mmol/L (126 mg/dL), and/or 5.7% ≤ HbA1c < 6.5%.
  2. Hypertension: Medically documented history of hypertension, or newly diagnosis of hypertension at screening (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg, measured at least 3 times on different days).
  3. Dyslipidemia: Medically documented history of dyslipidemia (with or without medication), or at screening TC ≥ 5.2 mmol/L (200 mg/dl), and/or LDL-C ≥ 3.4 mmol/L (130 mg/dl), and/or HDL-C < 1.0 mmol/L (40 mg/dl), and/or TG ≥ 1.7 mmol/L (150 mg/dl).
  4. Fatty liver disease: Evidence of fatty liver confirmed by imaging within 3 months prior to screening or newly diagnosed at screening.
  5. Obstructive sleep apnea syndrome.
  6. Complaint of weight-bearing joint pain (during or within 3 months prior to screening).
* Participants had a stable weight maintenance during the 3 months of dietary and physical activity prior to screening (participant-reported data acceptable) and no more than 5% weight fluctuation, which is calculated as: (maximum weight - minimum weight during the 3 months of dietary and exercise control prior to screening)/maximum weight *100%.
* Female participants of childbearing potential (including female partners of male participants) who have no plans to father a child or donate sperm from screening until 6 months after the last dose, and are willing to use at least one effective contraception.
* Participants who well understand the study objectives, can communicate well with the investigator and to understand and comply with the requirements of this study, such as following the protocol medication and lifestyle intervention.

Exclusion Criteria:

* Obesity secondary to underlying medical conditions or drug therapy, including but not limited to hypercortisolism (e.g., Cushing's syndrome), polycystic ovary syndrome, or obesity due to pituitary/hypothalamic damage; OR weight increase attributable to elevated non-fat mass (e.g., edema) at screening or randomization.
* Have diabetes mellitus (including type 1 diabetes, type 2 diabetes, diabetes secondary to pancreatic injury, or other types of diabetes) or diagnosed with type 2 diabetes at screening/randomization, defined as HbA1c ≥ 6.5%, and/or fasting plasma glucose ≥ 7.0 mmol/L (126 mg/dL), and/or random plasma glucose ≥ 11.1 mmol/L (200 mg/dL).
* One or more episodes of unexplained hypoglycemic events within 3 months prior to screening, defined as FPG < 2.8 mmol/L (50 mg/dL) and/or presence of clinically significant hypoglycemic symptoms (symptoms of sympathetic activation [e.g., palpitations, anxiety, sweating, dizziness, hand tremble, hunger, etc.] and neuroglycopenic symptoms [e.g., altered consciousness, cognitive impairment, convulsions, and coma]).
* History of psychiatric disorders, addictive disorders, or other conditions that may compromise the subject's ability to provide informed consent; OR history of unstable anxiety and/or depression that, in the investigator's judgment, remains clinically significant.
* Have any lifetime history of a suicidal attempt or suicidal behavior.
* History of major cardiovascular or cerebrovascular disease within 6 months prior to screening, defined as:

  1. Acute myocardial infarction (MI), percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), heart valve repair/replacement, unstable angina, hemorrhagic stroke (stroke), ischemic stroke (including transient ischemic attack [TIA]).
  2. Congestive heart failure of New York Heart Association (NYHA) class III or IV.
* History of cardiac arrhythmias, including torsades de pointes, ventricular tachycardia, or second- or third-degree atrioventricular block.
* Have a family or personal history of long QT syndrome, or family history of sudden death in first-degree relatives (parent, child, sibling) before the age of 40 years, and/or personal history of unexplained syncope within 1 year prior to screening.
* History of gout within 6 months prior to screening.
* History of proliferative retinal disease or maculopathy.
* History of malignancy within 5 years prior to screening (except cured basal cell carcinoma of skin and cervical carcinoma in situ) or newly diagnosed malignancy at screening.
* Have a family or personal history (parents, children, and siblings) of medullary thyroid cancer (MTC) or Multiple Endocrine Neoplasia Syndrome Type 2 (MEN2).
* Abnormal thyroid function tests at screening (thyroid-stimulating hormone [TSH] > 6 mIU/L or < 0.4 mIU/L) not adequately controlled by stable medication doses (defined as stable dosage for ≥3 months), untreated subclinical hypothyroidism (TSH <10.0 mIU/L with normal free T3 [FT3] and free T4 [FT4] levels) is permitted.
* History of significant gastrointestinal disease (e.g., active ulcer) or gastrointestinal surgery (except appendectomy, cholecystectomy, or other gastrointestinal endoscopic procedures judged by the investigator as having no significant effect on gastrointestinal motility) or clinically significant gastric emptying abnormality (e.g., pyloric obstruction, gastroparesis) within 6 months prior to screening.
* History of gastrointestinal disorders (e.g., chronic diarrhea, constipation, hemorrhoidal bleeding-whether resolved or not) deemed clinically significant by the investigator, OR acute exacerbation of hemorrhoids within 3 months prior to screening.
* History of acute or chronic pancreatitis, or serum amylase or lipase > 1.5 × upper limit of normal (ULN) at screening.
* Previous acute or chronic hepatitis, or symptoms and signs of any other liver disease other than non-alcoholic fatty liver disease, or any of the following, as determined by laboratory tests at screening:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 × ULN.
  2. Blood total bilirubin (TBIL) ≥ 1.5 × ULN.
  3. Alkaline phosphatase (ALP) ≥ 3 × ULN.
* Symptomatic cholecystitis or biliary diseases within 1 year prior to screening, except those with documented resolution of biliary stones following treatment.
* Hypersensitivity or suspected hypersensitivity to glucagon-like peptide 1 receptor agonist (GLP-1RA) drugs or excipients.
* History of drug abuse or dependence prior to screening.
* High alcohol consumption within 3 months prior to screening (defined as an average daily consumption of more than 25 g of pure alcohol [equivalent to 750 mL of beer or 250 mL of wine or 50 g of liquor]).
* Have current or history of treatment with medications that may cause significant weight gain within 3 months prior to screening, including but not limited to:

  1. Approved/unapproved marketed weight-loss drugs: orlistat, sibutramine hydrochloride, phentermine, phentermine-topiramate, naltrexone-amfebutamone, tirzepatide, semaglutide, liraglutide, beinaglutide, phendimetrazine, methylamphetamine, etc.
  2. Glucagon-like peptide 1 receptor (GLP-1R) agonists or GLP-1R/glucagon receptor (GCGR) agonists or glucose-dependent insulinotropic polypeptide receptor (GIPR)/GLP-1R agonists or GIPR/GLP-1R/GCGR agonists or dipeptidyl peptidase 4 (DPP-4) inhibitors.
* History of bariatric surgery (excluding acupuncture/cupping/catgut embedding for bariatric surgery, liposuction, and abdominoplasty performed >1 year prior to screening) or plans to undergo bariatric surgery or acupuncture/cupping/catgut embedding, liposuction, abdominoplasty during the study period.
* Symptomatic cholecystitis or biliary diseases within 1 year prior to screening, except those with documented resolution of biliary stones following treatment.
* Major or medium-sized surgery, or severe trauma or serious infection within 3 months prior to screening, which, as assessed by the investigator, would preclude trial participation, or planned surgery during the study period (excluding outpatient procedures deemed by the investigator to have no impact on subject safety or trial outcomes).
* History of organ transplant.
* Use of any drug or food known to potently or moderately inhibit or induce cytochrome P450 3A4 enzyme (CYP3A4) and/or inhibit P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study.
* Uncontrolled hypertension at screening, defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg (verified prior to randomization. Blood pressure measurement should be performed after ≥5 minutes of seated rest, initial measurement followed by a second measurement after ≥1 minute, the final value will be the arithmetic mean of the two measurements (rounded to the nearest integer). If the difference between the first two measurements is ≥5 mmHg for either SBP or DBP, a third measurement shall be taken after ≥1 minute, the final value will be the arithmetic mean of all three measurements (rounded to the nearest integer).
* Positive hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody or syphilis antibody at screening.
* If any of the following laboratory abnormalities are present at screening:

  1. Blood calcitonin ≥ 50 ng/L.
  2. Estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73 m2, calculated according to the CKD-EPI formula, as shown in Appendix VIII.
  3. Poorly controlled severe dyslipidemia with TG ≥ 5.65 mmol/L (500 mg/dL) despite the use of conventional lipid-lowering drugs.
  4. Prothrombin time-international normalized ratio (INR) > 1.5 × ULN.
  5. Hemoglobin < 110 g/L (female) or < 120 g/L (male).
* QTcF > 450 ms for male or QTcF > 470 ms for female at screening, measured after rest at least 5 min (repeat the measurement once and take the mean value [rounded off to integer]; the interval between measurements is 2 min±60 s).
* Currently participating in any other clinical study, or if received any investigational product or medical devices within ≤ 3 months or 5 half-lives (t1/2) prior to screening, whichever is longer.
* Donation or loss of ≥ 400 mL of blood or transfusion within 3 months prior to screening.
* Female participants during pregnancy or lactation.
* The investigator, site personnel, and/or their immediate family members directly related to the study. An immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Participants who may be unable to complete this study for other reasons, or have other conditions that, as assessed by the investigator, will make the participant unsuitable for participation in this study, for example, the participant refuses to use only the weight-loss drugs specified in the protocol during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-09 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Body Weight From Baseline at Week 12 | Baseline, Week 12
  Percent Change in Body Weight From Baseline at Week 12

SECONDARY OUTCOMES:
Change in Body Weight (kg) from Baseline at Week 12 | Baseline, Week 12
Percentage of Study Participants Who Achieve ≥5% and ≥10% Body Weight Reduction at Week 12 | Baseline, Week 12
Change in BMI (kg/m2) from Baseline at Week 12 | Baseline, Week 12
Change in Waist Circumference from Baseline at Week 12 | Baseline, Week 12
Change in hyperlipidemia (TC, TG, LDL-C, HDL-C, nHDL-C) From Baseline at Week 12 | Baseline, Week 12
Change in Blood Pressure (SBP, DBP) from Baseline at Week 12 | Baseline, Week 12
Change in Blood Glucose (HbA1c, FPG) from baseline at Week 12 | Baseline, Week 12
Collect the incidence of adverse events (AEs) through vital signs, physical examination, laboratory tests, 12-lead electrocardiogram, etc. | Baseline, Week 13

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Ch’ang-ch’un, Jilin, China

IPD SHARING:
Plan to Share IPD: No